CLINICAL TRIAL: NCT05811078
Title: The Effect of Education Including Peer Interactive Group Support on Metabolic Control ın Adolescents wıth Type One Diabetes a Randomized Controlled Study
Brief Title: Metabolic Control Adolescents Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toros University (Other)
Responsible Party: Principal Investigator, Didem Polat Kulcu, principle ınvestigator, Toros University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: TorosU
Record Dates: First submitted 2022-10-07; First posted 2023-04-13 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: 13-18 Year; Diagnosed at Least 6 Months Ago; HbA1C> 7.5; Being Able to Read and Write
Keywords: Type 1 diabetes; metabolic control; adolescence; nursing
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: randomized controlling trail
Who Masked: Participant
Masking Description: Adolescents who met the inclusion criteria of the study were listed and their names were written to someone who was not involved in the study. The adolescents included in the list formed by this person who was excluded from the study were randomly assigned to the experimental and control groups according to the block randomization method in order to eliminate the selection bias and to ensure the balance in the number of individuals between the groups. From here, all possible possibilities were created and the blocks were arranged so that there were 4 individuals (2 experiments, 2 controls) in each block. Each block was given a number and the assignment was made using the https://www.randomizer.org/ address.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enterprise Group (Experimental): The contents of the research were created according to the Roy Adaptation model. Each session lasted an average of 2 hours.
  Peer interactive group support sessions were administered to the adolescents in the intervention group, one week apart. There were 7 sessions in total. The sitting arrangement of the training room is designed to allow children to interact with each other . The sessions lasted an average of 90 minutes as two 45-minute sessions. Between sessions, breaks that lasted for about 15 minutes were given and refreshments prepared for individuals with Type 1 diabetes were served during the breaks. During the break, the adolescents were given the opportunity to interact with each other by chatting. Fun exercise and kitchen workshop activities were also organized as interaction sessions in the initiative group.
  Interventions: Behavioral: training sessions with peer interactive group
- Control Group (No Intervention): Adolescents and their families were informed in the diabetes education room in the pediatric endocrine service of the hospital where the study was conducted, and their written consent was obtained. Within the scope of the pre-test, "Diabetes Adolescent Diagnosis Form", "Diabetes Information Evaluation Form", "Diabetes Management Self-Efficacy Scale in Adolescents with Type 1 Diabetes" and "Child's Attitude towards Own Disease Scale" were applied. Then, individual diabetes education was given by the diabetes education nurse as a hospital routine. Three months after the training, the adolescents were called by phone to the hospital for control, HbA1c follow-up was taken and post-test applications were made.

INTERVENTIONS:
Behavioral: training sessions with peer interactive group — Data were collected with data collection forms consisting of " Diabetes Adolescent Diagnosis Form", "Diabetes Information Evaluation Form", "Diabetes Management Self-Efficacy Scale in Adolescents with Type 1 Diabetes" and "Child's Attitude towards Own Disease Scale" .
  Arms: Enterprise Group

SUMMARY:
Purpose of the research; The aim of this study is to examine the effect of education including peer-interactive group support to be given to adolescents diagnosed with Type 1 diabetes with poor glycemic control in the 13-18 age group on metabolic control of adolescents.

DETAILED DESCRIPTION:
The lack of a certificate program specific to pediatric diabetes nursing of the Ministry of Health in our country and the insufficient number of diabetes education nurses show that the pediatric population is not adequately trained to provide diabetes management. Along with these obstacles, the lack of use of an evidence-based standard education program reveals the need for effective intervention programs that include approaches specific to adolescents, who are a particularly risky group. Peer interaction can be used as an effective approach to increase adolescents' adherence to treatment. Thus, adolescents who isolate themselves are given the opportunity to cope with the disease and to share with other children. It has been determined that there is no study in the literature that includes peer-interactive group support on adolescents with a diagnosis of Type 1 diabetes who have poor glycemic control but have repeated hospitalizations. This situation shows that there is a need for a study to evaluate the effect of educational intervention including peer-interactive group support on repeated hospitalizations in adolescents with Type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* be between 13-18 years old
* Diagnosed at least 6 months ago
* HbA1C level > 7.5
* Having repeated hospitalizations at least twice
* Living in Mersin city center
* Being able to communicate in Turkish
* Being able to read and write

Exclusion Criteria:

* - Using an insulin pump
* Having a chronic disease other than diabetes,
* Diseases that affect cognitive functions, hearing and vision impairments

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Implementation of trainings containing peer interactive group support to adolescents and application of scales | 7 weeks
  The contents of the research were created according to the Roy Adaptation model. Each session lasted an average of 2 hours.
  Peer interactive group support sessions were administered to the adolescents in the intervention group, one week apart. There were 7 sessions in total. The sessions lasted an average of 90 minutes as two 45-minute sessions. Between sessions, breaks that lasted for about 15 minutes were given and refreshments prepared for individuals with Type 1 diabetes were served during the breaks. During the break, the adolescents were given the opportunity to interact with each other by chatting. Fun exercise and kitchen workshop activities were also organized as interaction sessions in the initiative group.

SECONDARY OUTCOMES:
Evaluation of Data | one year
  The data obtained from the research were evaluated using appropriate statistical methods. In the analysis of comparative data, parametric or nonparametric tests were used by evaluating the conformity to the normal distribution . As descriptive statistics; numbers and percentages are given. In addition, mean and standard deviation values are given for those with normal distribution, and minimum and maximum values, median and percentiles of 25-75 % for those who do not show normal distribution.

CONTACTS AND LOCATIONS:
Locations (1):
- Toros Üniversty, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
may be shared upon reasonable request from the author
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2024
Access Criteria: may be shared upon reasonable request from the author